CLINICAL TRIAL: NCT02561988
Title: A Phase 1 Study of BLU-285 in Patients With Advanced Systemic Mastocytosis (AdvSM) and Relapsed or Refractory Myeloid Malignancies
Brief Title: (EXPLORER) Study of BLU-285 in Patients With Advanced Systemic Mastocytosis (AdvSM) and Relapsed or Refractory Myeloid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLU-285-2101; 2015-001661-12 (EudraCT Number)
Record Dates: First submitted 2015-09-15; First posted 2015-09-29 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Aggressive Systemic Mastocytosis; Systemic Mastocytosis-associated Hematologic Non-mast Cell Disease; Mast Cell Leukemia; Relapsed or Refractory Myeloid Malignancies
MeSH Terms: conditions — Mastocytosis, Systemic; Leukemia, Mast-Cell; Recurrence | interventions — avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avapritinib (also known as BLU-285) (Experimental): Avapritinib tablets for oral administration. Avapritinib will be dosed daily for 28 day cycles.
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib

SUMMARY:
This is a Phase 1, open-label, dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and antineoplastic activity of avapritinib (also known as BLU-285), administered orally (PO), in adult patients with advanced systemic mastocytosis and other relapsed or refractory myeloid malignancies. The study consists of 2 parts:, dose-escalation (Part 1) and expansion (Part 2).

ELIGIBILITY:
Inclusion Criteria:

For Part 1:Patients must have one of the following diagnoses based on World Heath Organization (WHO) diagnostic criteria:

* Aggressive systemic mastocytosis (ASM).
* Systemic mastocytosis with an associated hematologic neoplasm (SM-AHN) and at least 1 C-finding attributable to systemic mastocytosis (SM). The AHN must be myeloid, with the following exceptions that are excluded: Acute myeloid leukemia (AML), Myelodysplastic syndrome (MDS) that is very high- or high-risk as defined by the International prognostic scoring system for myelodysplastic syndromes (IPSS-R) and Philadelphia chromosome positive malignancies.
* Mast cell leukemia (MCL).
* Histologically- or cytologically- confirmed myeloid malignancy that is relapsed or refractory to standard treatments. AML, MDS that is very high- or high-risk as defined by the IPSS-R, and Philadelphia chromosome positive malignancies are excluded.
* Upon discussion with the sponsor, other relapsed or refractory, potentially avapritinib-responsive hematologic neoplasms (e.g., evidence of aberrant KIT or platelet derived growth factor receptor (PDGFR) signaling) may be considered for enrollment.

For Part 2, patients must have one of the following diagnoses, based on WHO diagnostic criteria:

* ASM.
* SM-AHN. The AHN must be myeloid, with the following exceptions that are excluded: AML, MDS that is very high- or high-risk as defined by the IPSS-R, and Philadelphia chromosome positive malignancies.
* MCL.

For Part 2, Cohort 2, patients must have at least 1 measurable C-finding per modified IWG-MRT-ECNM criteria at Baseline, attributed to SM unless diagnosis is MCL, which does not require a C-finding.

* Cytopenias: ANC < 1.0 × 10⁹/L or hemoglobin < 10 g/dL or platelet count < 75 × 10⁹/L.
* Symptomatic ascites or pleural effusion requiring medical intervention such as: use of diuretics (Grade 2) or ≥ 2 therapeutic paracenteses or thoracenteses (Grade 3) at least 28 days apart over the 12 weeks before study entry and 1 of the procedures is performed during the 6 weeks before study start (C1D1).
* ≥ Grade 2 abnormalities in direct bilirubin (> 1.5 × upper limit of normal [ULN]), aspartate aminotransferase (AST; > 3.0 × ULN), alanine aminotransferase (ALT; > 3.0 × ULN), or alkaline phosphatase (> 2.5 × ULN) with 1 of the following present: ascites or clinically relevant portal hypertension or liver mast cell infiltration that is biopsy-proven or no other identified cause of abnormal liver function.
* ≥ Grade 2 hypoalbuminemia (< 3.0 g/dL).
* A spleen that is palpable ≥ 5 cm below the left costal margin.
* Transfusion-dependent anemia defined as: transfusion of ≥ 6 units packed red blood cells (PRBCs) in the 12 weeks before start of treatment (C1D1) and most recent transfusion occurring during the preceding 4 weeks and transfusion administered for hemoglobin ≤ 8.5 g/dL and reason for transfusion is not bleeding, hemolysis, or therapy-related.

Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.

Exclusion Criteria:

* QT interval corrected using Fridericia's formula (QTcF) >480 milliseconds
* Platelet count <50,000/μL (within 4 weeks of the first dose of study drug) or receiving platelet transfusion(s)
* Absolute neutrophil count <500/μL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >3 x the upper limit of normal (ULN); >5 × ULN if associated with clinically suspected liver infiltration by mastocytosis or another disease for which the patient enrolled into the study
* Total bilirubin >1.5 × ULN; >3 × ULN if associated with liver infiltration by the disease being treated or in the presence of Gilbert's Disease (In the case of Gilbert's disease, a direct bilirubin > 2.0 ULN would be an exclusion.)
* Estimated (Cockroft-Gault formula) or measured creatinine clearance <40 mL/min
* Brain malignancy or metastases to the brain
* History of a seizure disorder or requirement for anti-seizure medication
* Known risk of intracranial bleeding, such as a brain aneurysm or history of subdural or subarachnoid bleeding
* Eosinophilia and known positivity for the FIP1L1-PGDFRA fusion, unless the patient has demonstrated relapse or progressive disease on prior imatinib therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of avapritinib (also known as BLU-285) | During cycle 1 (28 days) of treatment
Number of patients with adverse and serious adverse events and changes in physical findings, vital signs, clinical laboratory results and ECG findings | Approximately 24 months
Recommended Phase 2 dose (RP2D) of avapritinib | Approximately 24 months

SECONDARY OUTCOMES:
Maximum plasma concentration of avapritinib | Every cycle (28 days) up to cycle 4
  Blood samples may be taken at pre-dose, and 0.5, 1, 2, 4, 8 and 24 hrs post dose (plus 10 and 48 hrs post dose in Part 2) on Cycle 1 Day 1 and Cycle 1 Day 15, Pre-dose of Cycle 2 to 4, Day 1
Time to maximum plasma concentration of avapritinib | Every cycle (28 days) up to cycle 4
  Blood samples may be taken at pre-dose, and 0.5, 1, 2, 4, 8 and 24 hrs post dose (plus 10 and 48 hrs post dose in Part 2) on Cycle 1 Day 1 and Cycle 1 Day 15, Pre-dose of Cycle 2 to 4, Day 1
Overall Response Rate | 8, 24, 40, 68 and every 24 weeks until patient terminates from the study (approximately 24 months)
  Including complete remission (CR), CR with partial recovery of peripheral blood (CRh), partial remission (PR) and clinical improvement (CI) using modified International Working Group Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European competence network on mastocytosis (ECNM) criteria; and duration of response (DOR)
Morphologic response | ≥ 12 weeks
  Including morphologic complete remission (mCR), morphologic CR with partial recovery of peripheral blood (mCRh), and morphologic partial remission (mPR) based on Pure Pathologic Response
Changes in levels of serum tryptase and levels of V-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog (KIT) D816V allele burden in blood | Cycle (C)1Day (D)1, C1D15, C2D1, C3D1, C5D1, C7D1, C11D1, C18D1 every 6 cycles thereafter and at disease progression. (approximately 24 months)
Changes in patient reported symptoms and quality of life using the Patient Global Impression of Symptom Severity (PGIS) scale | Part 2 only - Day 1 of Cycles 1-12
  Defined as change from Baseline
Changes in patient reported quality of life using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C-30) | Part 2 only - Day 1 of Cycles 1-12
  Defined as change from Baseline
Changes in patient reported outcomes using the advanced SM symptom assessment form (AdvSM-SAF) | Part 2 only - daily from Day -7 through Cycle 12
  Defined as change from Baseline
Change in liver volume by imaging | Day 1 of Cycles 5-18, and every 6 cycles thereafter (each cycle is 28 days)
  mL
Change in spleen volume by imaging | Day 1 of Cycles 5-18, and every 6 cycles thereafter (each cycle is 28 days)
  mL

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - Stanford Cancer Institute, Stanford, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mount Sinai Hospital, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- United Kingdom (2):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guy's Hospital, London

REFERENCES:
- [Derived] Reiter A, Gotlib J, Alvarez-Twose I, Radia DH, Lubke J, Bobbili PJ, Wang A, Norregaard C, Dimitrijevic S, Sullivan E, Louie-Gao M, Schwaab J, Galinsky IA, Perkins C, Sperr WR, Sriskandarajah P, Chin A, Sendhil SR, Duh MS, Valent P, DeAngelo DJ. Efficacy of avapritinib versus best available therapy in the treatment of advanced systemic mastocytosis. Leukemia. 2022 Aug;36(8):2108-2120. doi: 10.1038/s41375-022-01615-z. Epub 2022 Jul 5. PMID 35790816
- [Derived] Reiter A, Schwaab J, DeAngelo DJ, Gotlib J, Deininger MW, Pettit KM, Alvarez-Twose I, Vannucchi AM, Panse J, Platzbecker U, Hermine O, Dybedal I, Lin HM, Rylova SN, Ehlert K, Dimitrijevic S, Radia DH. Efficacy and safety of avapritinib in previously treated patients with advanced systemic mastocytosis. Blood Adv. 2022 Nov 8;6(21):5750-5762. doi: 10.1182/bloodadvances.2022007539. PMID 35640224
- [Derived] DeAngelo DJ, Radia DH, George TI, Robinson WA, Quiery AT, Drummond MW, Bose P, Hexner EO, Winton EF, Horny HP, Tugnait M, Schmidt-Kittler O, Evans EK, Lin HM, Mar BG, Verstovsek S, Deininger MW, Gotlib J. Safety and efficacy of avapritinib in advanced systemic mastocytosis: the phase 1 EXPLORER trial. Nat Med. 2021 Dec;27(12):2183-2191. doi: 10.1038/s41591-021-01538-9. Epub 2021 Dec 6. PMID 34873347